CLINICAL TRIAL: NCT06926478
Title: Clinical Trial to Evaluate Short-term Safety of Subconjunctival Adalimumab in Combination With Type 1 Boston Keratoprosthesis Implantation
Brief Title: Subconjunctival Humira for Boston Keratoprosthesis
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Massachusetts Eye and Ear Infirmary (Other)
Responsible Party: Principal Investigator, Thomas H. Dohlman, MD, Principal Investigator, Massachusetts Eye and Ear Infirmary
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025P000846
Record Dates: First submitted 2025-03-25; First posted 2025-04-13 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2025-04

CONDITIONS: Penetrating Keratoplasty; Multiple Graft Failure; Ocular Cicatricial Pemphigoid; Stevens-Johnson Syndrome
Keywords: Kpro; Boston Kpro; Keratoprosthesis; Type-1 Boston Kpro
MeSH Terms: conditions — Pemphigoid, Benign Mucous Membrane; Stevens-Johnson Syndrome | interventions — Adalimumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Adalimumab (Humira) (Experimental): This arm will receive the study intervention.
  Interventions: Drug: Adalimumab Injection

INTERVENTIONS:
Drug: Adalimumab Injection — 10% (4.0mg/0.04ml) dissolved in sterile saline to be injected once during the time of the Boston Keratoprosthesis (Kpro) Surgery.
  Other Names: Humira

SUMMARY:
This trial is studying the safety and tolerability of receiving an injection of adalimumab (Humira) during the Boston Keratoprosthesis (KPro) surgery.

DETAILED DESCRIPTION:
This is a Phase I, Open-label, IND trial for participants undergoing a Boston Keratoprosthesis (KPro) procedure, to receive an injection of adalimumab (Humira), to study the safety and tolerability as well, to study whether there is a decrease to post surgical complications, and symptoms that participants would experience, if they did not receive the injection.

The study will recruit eight (8) participants, who will be monitored for thirty (30) days after the surgery, through eye examination and eye photos.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Individuals eligible for keratoprosthesis surgery, as determined by standard-of-care eligibility criteria
* Patients with poor prognosis for corneal transplantation, severe corneal opacity and/or vascularization
* Patients with vision worse than 20/200 in the eligible eye, and contralateral eye with vision less than 20/40
* Patients with intact nasal light projection
* Willing and able to comply with study plan for the full duration of the study
* Willing and able to sign a written informed consent

Exclusion Criteria:

* Active tuberculosis or untreated latent tuberculosis (e.g., positive interferon-# release assay [IGRA] test, such as Quantiferon-gold)
* Untreated active hepatitis B or C infection.
* Ocular or periocular malignancy and/or infection
* Inability to wear contact lens
* Pregnancy (positive pregnancy test) or lactating
* Participation in another interventional study at the time of screening
* Any of the following baseline lab values

  1. White blood count <3500 cells per microliter
  2. Platelets <100,000 per microliter
  3. Hematocrit <30%
  4. AST or ALT >1.5X upper limit normal value
* Multiple sclerosis or other demyelinating disease
* Severe uncontrolled infection
* Moderate to severe heart failure (NYHA class III/IV)
* Active malignancy
* History of adalimumab intolerance
* Pregnancy or lactation
* Medical problems or drug or alcohol dependence problems sufficient to prevent adherence to treatment and study procedures.
* As judged by the investigator any patients that are questionable for their suitability in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2027-08-01 (Estimated); Study Completion 2028-08-01 (Estimated)

PRIMARY OUTCOMES:
Evaluation of Treatment Related Adverse Events. | 30 Days
  To evaluate safety following subconjunctival injection of adalimumab at the time of keratoprosthesis surgery in patients who have corneal problems of such severity that they require keratoprosthesis implantation. The incidence, severity, and duration of adverse events will be assessed and documented. Because the subjects in this study have corneal problems of such severity that they require keratoprosthesis implantation, special attention will be given to adverse events of particular concern, such as microbial keratitis, subconjunctival hemorrhage, subconjunctival inflammation, or retinal necrosis or retinal detachment

SECONDARY OUTCOMES:
Efficacy of adalimumab Injection though changes in visual acuity. | 30 Days
  This efficacy outcome measure will be analyzed though changes of any worsening of the best corrective visual acuity by 15 letters at every study visit.
Efficacy of adalimumab Injection though changes in Optic Nerve Cup-to-Disk Ratio | Every Two (2) Weeks After Implantation/Injection until Day 30
  This efficacy outcome measure will be analyzed through any changes to the cup-to-disk ratio. A normal ratio is 0.2mm
Efficacy of adalimumab Injection through incidences of Intraocular Inflammation | 30 Days
  This efficacy outcome measure will be analyzed though any incidences of intraocular inflammation that occurs post implantation/injection.
Efficacy of adalimumab Injection through changes in the Ocular Coherence Tomography (OCT) of the Optic Nerves | 30 Days
  This efficacy outcome measure will be analyzed though any changes in the retinal nerve fiber layer thickness (nerve edema).
Efficacy of adalimumab Injection though changes in the ocular coherence tomography (OCT) of the Retina | 30 Days
  This efficacy outcome measure will be analyzed though increases in the foveal retinal thicknesses by an increase of more than (>)100um in comparison to the previous study visit(s).

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Dohlman, MD, Principal Investigator — Massachusetts Eye and Ear
Locations (1):
- Massachusetts Eye and Ear, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No